CLINICAL TRIAL: NCT02604810
Title: An Open-label, Multi-center Study to Evaluate the Safety and Pharmacokinetics of IGSC 20% Administered for 6 Months in Subjects With Primary Immunodeficiency
Brief Title: Safety and Pharmacokinetics of IGSC 20% in Subjects With Primary Immunodeficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GTI1502
Record Dates: First submitted 2015-11-06; First posted 2015-11-13 (Estimated); Results first posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2018-09

CONDITIONS: Primary Immunodeficiency
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — Immunoglobulins; Caprylates; Chromatography; gamma-Globulins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IGIV-C 10% (Active Comparator): IV dose of Immune Globulin Injection (Human), 10% Caprylate/Chromatography Purified (Grifols)
  Interventions: Biological: IGIV-C 10%
- IGSC 20% (Experimental): Immune Globulin Subcutaneous (Human), 20% Caprylate/Chromatography Purified (Grifols)
  Interventions: Biological: IGSC 20%

INTERVENTIONS:
Biological: IGIV-C 10% — IGIV-C 10% infusions every 3 to 4 weeks based on previous IgG regimen
  Other Names: Immune Globulin Injection 10% Caprylate/Chromatography
  Arms: IGIV-C 10%
Biological: IGSC 20% — IGSC 20% weekly infusions with dose calculated based on previous IgG regimen
  Other Names: Immune Globulin Subcutaneous 20% Caprylate/Chromatography
  Arms: IGSC 20%

SUMMARY:
This study was designed to determine a dose of weekly subcutaneously administered Immune Globulin Subcutaneous (Human), 20% Caprylate/Chromatography Purified (Grifols) (IGSC 20%) that produces steady-state AUC of total IgG that was non-inferior to that of the regularly administered intravenous dose of Immune Globulin Injection (Human), 10% Caprylate/Chromatography Purified (Grifols) (IGIV-C 10%) in primary immunodeficiency subjects. This study was also designed to determine steady state trough total IgG levels after IGSC 20% infusion and after IGIV-C 10% infusion for comparison and to assess the safety and tolerability of IGSC 20%.

DETAILED DESCRIPTION:
This was a prospective, multi-center, open-label, single-sequence, 6-month, pharmacokinetic, safety and tolerability study of IGSC 20% in subjects with primary immunodeficiency. Approximately 50 subjects were to be enrolled in order to have approximately 30 adult subjects and 12 to 18 pediatric subjects (age 2-16 years) completing treatment with subcutaneously administered IGSC 20%.

This study included 3 treatment phases: Run-In Phase, IV Phase (IV administration of IGIV-C 10% treatment), and SC Phase (SC administration of IGSC 20%).

Subjects, depending on their current IgG treatment regimen, might be required to enter the Run-In Phase to receive IV IGIV-C 10% treatment (Sponsor provided) to achieve an approximately steady-state condition prior to entering the IV Phase. They then entered the IV Phase to determine the AUC profiles of IV infusions of IGIV-C 10%.

Subjects with a qualifying IV IGIV-C 10% treatment regimen (on stable IGIV-C 10% doses of 300-800 mg/kg) entered the IV Phase directly where they will receive IGIV-C 10%. In the IV Phase, steady-state IV PK assessments, including AUC, were to be performed.

After completing the IV Phase, subjects entered the SC Phase to receive weekly SC doses of IGSC 20% for at least 24 weeks.

The PK profiles of total IgG following administration of both IV (IGIV-C 10%) administration and SC (IGSC 20%) administration were determined and compared after reaching approximate steady-state conditions.

ELIGIBILITY:
Inclusion Criteria:

* Pre-existing diagnosis of primary immunodeficiency with features of hypogammaglobulinemia requiring IgG replacement therapy
* No serious bacterial infection within the last 3 months prior to or during Screening
* Currently on IgG replacement therapy (via IV or SC infusion) for ≥3 consecutive months. Subjects receiving IGIV must be receiving a dosage of 300 to 800 mg/kg per infusion
* Documented (at least once within previous 3 months) IgG trough level of ≥500 mg/dL on current IgG replacement therapy regimen

Exclusion Criteria:

* Known serious adverse reaction to immunoglobulin or any severe anaphylactic reaction to blood or any blood-derived product
* History of blistering skin disease, clinically significant thrombocytopenia, bleeding disorder, diffuse rash, recurrent skin infections, or other disorders where SC therapy would be contraindicated during the study
* Isolated IgG subclass deficiency, isolated specific antibody deficiency disorder, or transient hypogammaglobulinemia of infancy
* Nephrotic syndrome, and/or a history of acute renal failure and/or severe renal impairment, and/or on dialysis
* History (year prior to Screening or 2 episodes in lifetime ) of or current diagnosis of deep venous thrombosis or thromboembolism (eg, deep vein thrombosis, myocardial infarction, cerebrovascular accident or transient ischemic attack)
* Acquired medical condition known to cause secondary immune deficiency, such as chronic lymphocytic leukemia, lymphoma, multiple myeloma, chronic or recurrent neutropenia (absolute neutrophil count less than 1000/μL [1.0 x 10^9/L]), or human immunodeficiency virus infection/acquired immune deficiency syndrome
* Known previous infection with or clinical signs and symptoms consistent with current hepatitis B virus or hepatitis C virus infection
* Non-controlled arterial hypertension (systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg in adult subjects)
* Receiving any of the following medications: (a) immunosuppressants including chemotherapeutic agents, (b) immunomodulators, (c) long-term systemic corticosteroids defined as daily dose >1 mg of prednisone equivalent/kg/day for>30 days Note: Intermittent courses of corticosteroids of not more than 10 days would not exclude a subject. Inhaled or topical corticosteroids are allowed.

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (20):
  - UCLA Medical Center, Los Angeles, California
  - AIRE Medical of Los Angeles, Santa Monica, California
  - National Jewish Health, Denver, Colorado
  - University of Miami - Batchelor Children's Research Institute, Miami, Florida
  - Allergy Associates of The Palm Beaches, PA, North Palm Beach, Florida
  - University of South Florida, St. Petersburg, Florida
  - Emory Children's Center, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - The South Bend Clinic, South Bend, Indiana
  - Children's Hospital of Michigan - Wayne State University, Detroit, Michigan
  - Midwest Immunology, Plymouth, Minnesota
  - Washington University Medical Center, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Oklahoma Institute of Allergy and Asthma Clinical Research, Oklahoma City, Oklahoma
  - Vital Prospects Clinical Research Institute, PC, Tulsa, Oklahoma
  - Penn State University, Hershey, Pennsylvania
  - AARA Research Center, Dallas, Texas
  - Baylor Texas Children's Hospital, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Children's Hospital of Richmond at VCU, VCU Medical Center, Richmond, Virginia
- Canada (5):
  - Ottawa Hospital, Division of Infectious Disease and Respirology, Ottawa, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
  - McGill University Health Center, Montreal
  - Clinique d'asthme et d'allergie de Quebec, Québec
  - The Hospital for Sick Children, Toronto

REFERENCES:
- [Derived] Sleasman JW, Lumry WR, Hussain I, Wedner HJ, Harris JB, Courtney KL, Mondou E, Lin J, Stein MR. Immune globulin subcutaneous, human - klhw 20% for primary humoral immunodeficiency: an open-label, Phase III study. Immunotherapy. 2019 Nov;11(16):1371-1386. doi: 10.2217/imt-2019-0159. Epub 2019 Oct 17. PMID 31621458

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 61 subjects were screened for participation in this study. Of these 61 subjects, 8 subjects were considered screen failures. A total of 20 investigators in the United States enrolled subjects in this study. The first subject was enrolled in this study on 04 Jan 2016 and the date of the last subject's last study visit was 14 Dec 2017.
Pre-assignment Details: One subject was lost to follow-up before the IGIV-C Phase.
Groups:
- IGIV-C 10% First, IGSC 20% Second: IV dose of Immune Globulin Injection (Human), 10% Caprylate/Chromatography Purified (Grifols)
  IGIV-C 10%: IGIV-C 10% infusions every 3 to 4 weeks based on previous IgG regimen
  After completing the IGIV-C 10% infusions, subjects continued to receive IGSC 20% infusions.
  Immune Globulin Subcutaneous (Human), 20% Caprylate/Chromatography Purified (Grifols)
  IGSC 20%: IGSC 20% weekly infusions with dose calculated based on previous IgG regimen
Period: IGIV-C 10%, 4-5 Weeks
Arm/Group | IGIV-C 10% First, IGSC 20% Second
Started | 52
Completed | 49
Not Completed | 3
Period: IGSC 20%, 24 Weeks
Arm/Group | IGIV-C 10% First, IGSC 20% Second
Started | 49
Completed | 42
Not Completed | 7

BASELINE CHARACTERISTICS:
Population: Baseline data were collected for 53 enrolled subjects.
Arm/Group | IGIV-C 10% First, IGSC 20% Second
Number analyzed (Participants) | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15
  Between 18 and 65 years | 33
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (21.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 48
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 48
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: AUC in the IV Phase and SC Phases: Steady-state AUC of Total IgG Over a Regular Dosing Interval
Description: The primary PK endpoint (steady-state AUC values) analysis was performed using analysis of variance (ANOVA) using PK data from a total of 49 subjects from the IV phase and 39 subjects from the SC phase.
Time Frame: For intravenous infusion, predose, 0,1,3-16 hours and 1,2,3,5,7,14,21 or 28 days (2, 7, 21, or 28 days for pediatric subjects) post-dose and for subcutaneous infusion, pre-dose,1,3,4,5,7 days (3 and 7 days for pediatric subjects) post-dose
Population: The PK population consisted of all subjects who received study drugs and had sufficient and valid total IgG concentration versus time data for either the IV or SC Phase to allow calculation of AUC0-τ,SC or AUC0-τ,IV (the primary PK endpoint).
Measure: Geometric Mean (90% Confidence Interval); unit: h*mg/dL
Arm/Group | IGIV-C 10% | IGSC 20%
Number analyzed (Participants) | 49 | 39
h*mg/dL | 207921.5 [197865.8 to 218488.2] | 213141.4 [200568.6 to 226502.3]
Statistical Analysis 1: Comparison: IGIV-C 10% vs IGSC 20%; Test type: Non-Inferiority — Method of estimation = least-squares means based on analysis of variance (ANOVA) with a mixed-effect model. The lower bound of the 90% confidence interval (CI) for the geometric LSM ratio (SC/IV) of the primary PK endpoint of steady state AUC0-7 days for the PK population should be above 0.80; Geometric least-squares mean ratio = 1.04, 90% CI 2-sided [1.00 to 1.07]

2. Secondary Outcome: Mean Steady-state Trough (Pre-dose) Concentration of Total IgG Following IV Administration of IGIV-C 10% or SC Administration of IGSC 20%
Time Frame: For intravenous infusion, pre-dose at Week 1 and Week 3 or Week 4 and for subcutaneous infusion, predose at Weeks 13, 14, 17, and 21
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | IGIV-C 10% | IGSC 20%
Number analyzed (Participants) | 51 | 44
mg/dL | 957.13 [351.0 to 1920.0] | 1244.84 [651.5 to 2047.5]

ADVERSE EVENTS:
Time Frame: During the IV phase, the adverse event data were collected for 4 to 5 weeks. During the SC phase, the adverse event data were collected for 24 weeks.
Arm/Group | IGIV-C 10% | IGSC 20%
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/49
Serious Adverse Events (participants affected / at risk) | 1/52 | 2/49
Other Adverse Events (participants affected / at risk) | 6/52 | 35/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IGIV-C 10% (N=52) | IGSC 20% (N=49)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Intervertebral disc (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IGIV-C 10% (N=52) | IGSC 20% (N=49)
Sinusitis (Infections and infestations) | 3 (3) | 9 (10)
Infusion site bruising (General disorders) | 0 (0) | 3 (3)
Infusion site nodule (General disorders) | 0 (0) | 6 (9)
Infusion site pain (General disorders) | 0 (0) | 3 (3)
Bronchitis (Infections and infestations) | 2 (2) | 3 (3)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site may publish results from the Study, after providing Sponsor thirty days' notice prior to submitting a manuscript or other materials related to the Study to any outside party. At Sponsors' request, Site will remove any Confidential Information (other than Study results), and Site will upon Sponsors' request, delay publication or presentation for a period of up to one hundred twenty days to allow Sponsor to protect its interests in any Sponsor Inventions.

DOCUMENTS (2):
  • Study Protocol (2016-03-15): https://cdn.clinicaltrials.gov/large-docs/10/NCT02604810/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/10/NCT02604810/SAP_001.pdf